CLINICAL TRIAL: NCT07047118
Title: A Phase II, Randomized, Open-label, Multi-center Study of JSB462 (Luxdegalutamide) in Combination With Lutetium (177Lu) Vipivotide Tetraxetan in Adult Male Patients With PSMA-positive Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Study of JSB462 (Luxdegalutamide) Plus Lutetium (177Lu) Vipivotide Tetraxetan in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJSB462B12201; 2024-520155-24-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-05-20; First posted 2025-07-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Cancer, Castration-Resistant
Keywords: Prostate cancer; metastatic Castration Resistant Prostate Cancer (mCRPC); Castration-resistant; Prostate-Specific Membrane Antigen (PSMA); PSMA-positive; Radioligand Therapy (RLT); lutetium (177Lu) vipivotide tetraxetan; Phase 2; Open-label; Androgen Receptor Pathway Inhibitor (ARPI)
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): JSB462 100 mg QD + AAA617 7.4 GBq Q6W
  Interventions: Drug: JSB462; Drug: AAA617
- Arm 2 (Experimental): JSB462 300 mg QD + AAA617 7.4 GBq Q6W
  Interventions: Drug: JSB462; Drug: AAA617
- Arm 3 (Active Comparator): AAA617 7.4 GBq Q6W
  Interventions: Drug: AAA617

INTERVENTIONS:
Drug: JSB462 — Administered orally, daily and continuously (100 mg or 300 mg QD) until disease progression per PCWG3-modified RECIST v1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision
  Other Names: luxdegalutamide
  Arms: Arm 1; Arm 2
Drug: AAA617 — administered at 7.4 GBq intravenously every 6 weeks for up to 6 doses, unless there is disease progression per PCWG3-modified RECIST v1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision
  Other Names: Pluvicto; [177Lu]Lu-PSMA-617

SUMMARY:
This Phase II study aims to evaluate the efficacy and safety of the combination of JSB462 (also known as luxdegalutamide) at 100 mg and 300 mg QD doses + lutetium (177Lu) vipivotide tetraxetan (hereafter referred as AAA617) compared with AAA617 (control) in participants with metastatic Castration Resistant Prostate Cancer (mCRPC) with prior exposure to at least 1 Androgen Receptor Pathway Inhibitor (ARPI) and 0-2 taxane regimens and to select the recommended dose of the combination for phase III. Towards that end, the totality of the efficacy, safety, tolerability and pharmacokinetic (PK) data from participants randomized in the study will be evaluated.

DETAILED DESCRIPTION:
The study consists of a screening period, a randomization period, a treatment period, a post-treatment safety follow-up followed by a long-term follow-up period.

JSB462 administration starts at day 1 of randomization, whereas AAA617 administration starts at day 1 of treatment period. Participants in arm 1 and arm 2 will therefore receive JSB462 during the 14-day randomization period before first administration of AAA617.

* JSB462 is administered orally, daily and continuously (100 mg or 300 mg once a day (QD)) until disease progression per Prostate Cancer Working Group (PCWG) 3-modified Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision.
* AAA617 will be administered at 7.4 gigabecquerel (GBq) intravenously every 6 weeks for up to 6 doses, unless there is disease progression per PCWG3-modified RECIST v1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision.

During the post-treatment follow up period:

* Safety follow-Up: After discontinuation of study treatment, all participants will be followed for at least 1 safety follow-up visit (30 days [+/- 7 days] after end of treatment visit). Subsequent lines of therapy may be administered according to investigator's discretion after treatment discontinuation.
* Long-term follow-up: Starts after the Safety follow-up period and lasts until the end of study. Safety, efficacy and survival information may be collected from the participants during this period.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult male participants with histologically and/or cytologically confirmed adenocarcinoma of the prostate. Participants with mixed histology (neuroendocrine) are not eligible.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) grade ≤2.
* At least 1 bone or visceral metastatic lesion present on baseline CT, MRI, or bone scan imaging obtained ≤28 days prior to initiation of study treatment.
* Participants must be [68Ga]Ga-PSMA-11 PET/CT scan positive and eligible as determined by the sponsor's central reader.
* Participant must have prior exposure to at least one second generation ARPI in the metastatic/advanced setting.
* Previous treatment with a maximum of 2 taxane regimens is allowed.
* Participants eligible for PARPi and/or immune checkpoint inhibitor (per local testing and according to investigator's judgement) are eligible to participate if they have previous exposure to this(these) therapy(ies).

Key Exclusion Criteria:

* Prior treatment with any RLT (approved or investigational) is not allowed
* Prior treatment with a protein degrader compound that targets AR is not allowed

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-01-07 (Estimated); Study Completion 2028-11-04 (Estimated)

PRIMARY OUTCOMES:
Prostate Specific Antigen 50 (PSA50) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 30 months
  Prostate Specific Antigen 50 (PSA50) Rate is defined as the proportion of participants who achieve a ≥50% decrease from baseline at any timepoint, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between
Incidence rate of adverse events (AEs) | From date of randomization till 30 days safety fup, assessed up to approximately 30 months
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Number of participants with dose adjustments | From date of randomization till 30 days safety fup, assessed up to approximately 30 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) will be summarized by treatment arm.
Duration of exposure to study treatment | From date of randomization till 30 days safety fup, assessed up to approximately 30 months
  Dose interruptions, dose reductions, drug discontinuations, dose intensity, and duration of exposure to study treatment (all study drugs).

SECONDARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 41 months
  Radiographic Progression Free Survival (rPFS) is defined as the time between randomization and the first occurrence of disease progression (per PCWG3-modified RECIST 1.1 as assessed by the investigator) or death due to any cause
Overall Survival (OS) | From date of randomization until date of death from any cause, assessed up to approximately 41 months
  Overall Survival (OS) is defined as the time between randomization and death due to any cause
Incidence rate of adverse events (AEs) | From date of randomization until date of death from any cause, assessed up to approximately 41 months
  The analysis of adverse events and laboratory abnormalities will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Overall Response Rate (ORR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 41 months
  Overall Response Rate (ORR) is defined as the proportion of participants achieving a confirmed complete response (CR) or partial response (PR) per PCWG3-modified RECIST 1.1 as assessed by the investigator
Disease Control Rate (DCR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 41 months
  Disease Control Rate (DCR) is defined as the proportion of participants achieving a CR, PR or stable disease (SD) per PCWG3-modified RECIST 1.1 as assessed by the investigator
Duration of Response (DOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 41 months
  Duration of Response (DOR) is defined as the time between first documented CR/PR and disease progression or death due to any cause per PCWG3-modified RECIST 1.1 as assessed by the investigator
Time to Response (TTR) | From date of randomization until date of first documented Complete Response (CR) or Partial Response (PR), assessed up to approximately 41 months
  Time to response (TTR) is defined as the time from randomization to the date of first documented CR or PR per PCWG3-modified RECIST 1.1 as assessed by the investigator
Time to soft tissue progression (TTSTP) | From date of randomization until date of soft tissue radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 41 months
  Time to soft tissue progression (TTSTP) is defined as the time from randomization to the date of first documented radiographic soft tissue progression per PCWG3-modified RECIST 1.1 as assessed by the investigator
Prostate Specific Antigen 90 (PSA90) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 30 months
  Prostate Specific Antigen 90 (PSA90) Rate is defined as the proportion of participants who achieve a ≥90% decrease in PSA from baseline at any timepoint, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between.
Prostate Specific Antigen 30 (PSA30) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 30 months
  Prostate Specific Antigen 30 (PSA30) Rate is defined as the proportion of participants who achieve a ≥30% decrease from baseline at any timepoint, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between
Prostate Specific Antigen 0 (PSA0) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 30 months
  Prostate Specific Antigen 0 (PSA0) Rate is defined as the proportion of participants who achieve a PSA level <0.2 ng/ml at any timepoint after start of treatment, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between
Duration of biochemical response (DBR) | From date of date of first PSA50 response until date of PSA progression or death from any cause, assessed up to approximately 41 months
  Duration of biochemical response (DBR) is defined as the time between the first date of PSA50 response and the date of PSA progression (an increase ≥25% in PSA and an absolute increase of ≥2 ng/mL above the NADIR confirmed by a second value ≥3 weeks later if there is PSA decline from baseline, or a ≥25% increase and a ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline) or death due to any cause.
Time to first symptomatic skeletal event (TTSSE) | From randomization until the first occurrence of a new symptomatic bone fracture, spinal cord compression, tumor-related orthopedic surgery, radiation therapy for bone pain, or death, assessed up to 41 months.
  Time to first symptomatic skeletal event (TTSSE) is defined as the date of randomization to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first
Plasma concentrations of JSB462 and plasma concentrations of its metabolite ARV-767 | Day 1 of Cycles 1 and 2: Pre-dose/0hour and Post-dose 4hour +/- 1hour. Day 1 of Cycles 3 to 6: Pre-dose/0hour. End of Treatment Visit (EOT): through study treatment discontinuation, an average of 24 months. 1 cycle = 28 days.
  JSB462 pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels in JSB462 treatment arms.
Concentrations of AAA617 in blood over time and PK parameters from blood radioactivity data | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  AAA617 pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels in AAA617 treatment arm.
Area under the AAA617 concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of AAA617 | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf will be listed and summarized using descriptive statistics.
Observed maximum blood concentration (Cmax) of AAA617 | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Time of maximum observed blood concentration occurrence (Tmax) of AAA617 | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T1/2) of AAA617 | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-life will be listed and summarized using descriptive statistics.
Total systemic clearance for intravenous administration (CL) of AAA617 | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
Volume of distribution during the terminal phase following intravenous elimination (Vz) of AAA617 | Cycle 1: Day 1 (pre-dose/0hour, end of infusion (EOI), 1hour ±15minutes, 4hours ±30minutes), Day 2 (24hours ±2hours), Day 3 (48hours ±2hours), Day 8 (168hours ±12hours).Cycles 3 & 5: Day 1 (pre-dose/0hour, EOI), Day 3 (48hours ±2hours). 1 cycle=6 weeks.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz will be listed and summarized using descriptive statistics.
Radiation absorbed doses in organs and tumors for AAA617 | Cycle 1: Day 1 (1-4 hours), Day 2 (24 hours ±6 hours), Day 3 (48 hours ±6 hours), Day 8 (168 hours ±24 hours). Cycle 3: Day 1 (1-4 hours), Day 3 (48 hours ±6 hours). Cycle 5b (fit patients): Day 1 (1-4 hours), Day 3 (48 hours ±6 hours). 1 cycle=6 weeks.
  The organ absorbed radiation dose (Gy/GBq) as well as the effective radiation dose (mSv/GBq) will be evaluated and summarized descriptively.
Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | From date of randomization until date of death from any cause, assessed up to approximately 41 months
  The PRO-CTCAE is a patient-reported outcomes measurement system developed by the National Cancer Institute as a companion to the CTCAE. It includes items covering participant-reported symptomatic adverse events (AEs) from the CTCAE. Each symptomatic AE concept has up to three items evaluating frequency, severity, or interference, focused on the study population and treatment regimens.
  Participants respond on a 5-point scale for each item:
  * Frequency: Never, Rarely, Occasionally, Frequently, Almost constantly
  * Severity: None, Mild, Moderate, Severe, Very severe
  * Interference: Not at all, A little bit, Somewhat, Quite a bit, Very much
  The past 7-day recall version is used, focusing on relevant symptoms like fatigue, diarrhea, and hot flashes.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (10):
  - Cancer And Blood Spclsts of AZ, Casa Grande, Arizona
  - Providence Saint Johns Health Ctr, Santa Monica, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - XCancer Omaha LLC, Omaha, Nebraska
  - NYU Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Univ of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio, San Antonio, Texas
- Australia (3):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (3):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Beijing, China
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- France (3):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Tours
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Rostock
- Israel (6):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Roma, RM
- Netherlands (3):
  - Novartis Investigative Site, Nijmegen, Gerlderland
  - Novartis Investigative Site, Leeuwarden, Provincie Friesland
  - Novartis Investigative Site, Hoofddorp
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (4):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Seville
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com